CLINICAL TRIAL: NCT03715049
Title: Clinical Assessment of the Performance of a Fractional CO2 Laser System (Fraxel Repair Laser) Intended for Treatment of Perioral Rhytides/Wrinkles
Brief Title: Fractional CO2 Laser System (Fraxel Repair Laser) Intended for Treatment of Perioral Rhytides/Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fraxel Laser for Upper Lip
Record Dates: First submitted 2014-04-30; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Wrinkle
Keywords: upper lip wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fraxel Laser Treatment (Other): Using the energy and density settings within the FDA approved limits (5-40mJ at 30-100% density) that were narrowed down by the pre-clinical portion of the study, and analysis of abdominal and facial tissue treated in Objective 1, up to thirty (30) subjects will be recruited and treated one (1) time in the perioral region of the upper lip and followed for 6 months (study design below). The acute effects of the laser application will be determined by subjective analysis using the wrinkle severity scores.
  Interventions: Procedure: Fraxel Laser Treatment

INTERVENTIONS:
Procedure: Fraxel Laser Treatment — The device to be used in this study is a FDA approved device [510(k) approval] used for aesthetic dermatological procedures. The Fraxel Repair laser system utilizes a sealed off, all metal carbon dioxide gas tube that is radio frequency (RF) excited and air cooled, emitting light at a wavelength of 10.6 μm with programmable pulse duration and frequency. The Fraxel Repair laser has a continuous motion (rolling) optical tracking system. The Fraxel system consists of a treatment component and an internal control component. The treatment component consists of the laser delivery handpiece. A computer with a touch screen keyboard to enter subjects' information also provides controls for the fractionated delivery of the 10.6 μm beam.

SUMMARY:
Objective 1: To evaluate the effect and histologic (cellular) changes associated with varying energy and density settings of the Fraxel Repair Laser to determine an optimal dose response.

Objective 2: To evaluate the clinical response associated with variable energy and density settings of fraxel laser treatment in the upper lip. Overall assessment of clinical outcome and safety will be based clinic visits and evaluation of pre- and post- procedural photos. The subject's assessment of satisfaction will be characterized using a non-parametric assessment scale at each follow-up period.

DETAILED DESCRIPTION:
To evaluate the clinical response associated with variable energy and density settings of fraxel laser treatment in the upper lip. Overall assessment of clinical outcome and safety will be based clinic visits and evaluation of pre- and post- procedural photos. The subject's assessment of satisfaction will be characterized using a non-parametric assessment scale at each follow-up period.

This is a multi-site, non-randomized, non-controlled investigator initiated study designed to follow a total of 30 qualified and consenting subjects treated with one Fraxel Repair treatment in the course of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18-75 years of age.
* Subjects who can read, understand, and sign the Informed Consent Form.
* Subjects willing and able to comply with all study requirements.
* Fitzpatrick skin type I-IV (Although the systems are cleared for all skin types I- VI, it is recommended to use the Matrix applicators on skin types I- V).

Exclusion Criteria:

* Subjects with active localized or systemic infections.
* Immunocompromised subjects.
* Subjects with coagulation disorder.
* History of skin photo sensitivity disorders, or use of photosensitizing drugs (e.g., tetracycline or sulfa drugs).
* Pregnant and/or lactating (All female volunteers will be advised about using birth control during the period of study).
* In the opinion of the trained clinician, subject is unwilling or unable to adhere to all study requirements, including application and follow-up visits.
* Use of Accutane® within the past 6 months.
* Subjects with a history of radiation therapy to the treatment area.
* Subject has a history of allergy to lidocaine or ester-based local anesthetics.
* Subjects with any skin pathology or condition that could interfere with evaluation or with the use of typical ancillary medical treatments or care used before, during or after treatments.
* Subjects have undergone dermatological procedures (e.g., laser or light treatments) for the treatment of wrinkles, skin resurfacing, or skin rejuvenation in the treatment area within 1 year of study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in the lip wrinkles from baseline to 1 month | 1 month
  The primary outcome measure of effectiveness will be a paired comparison of baseline to 1, 3, and 6 month follow-up ratings for wrinkles using a Merz Aesthetic Lip Line score (0 none 1-4). Safety will be defined as an absence of hypopigmentary changes and by a restoration of hyperpigmentary changes to mild or less at 1 month. Photographs of treated skin at follow-up visits will be compared to baseline to document the healing time course and may be used for blinded scoring evaluations (0-9 scales) of wrinkles, skin texture and color changes. The investigator will grade the epidermal response including side effects and adverse events using the 0 to 10 grading scale.
Change in lip wrinkle from baseline to 3 months | 3 month
  The primary outcome measure of effectiveness will be a paired comparison of baseline to 3 months ratings for wrinkles using a Merz Aesthetic Lip Line score (0 none 1-4). Safety will be defined as an absence of hypopigmentary changes and by a restoration of hyperpigmentary changes to mild or less at 3 month. Photographs of treated skin at follow-up visits will be compared to baseline to document the healing time course and may be used for blinded scoring evaluations (0-9 scales) of wrinkles, skin texture and color changes. The investigator will grade the epidermal response including side effects and adverse events using the 0 to 10 grading scale.
Change in the lip wrinkles from baseline to 6 month | 6 month
  The primary outcome measure of effectiveness will be a paired comparison of baseline to 6 month follow-up ratings for wrinkles using a Merz Aesthetic Lip Line score (0 none 1-4). Safety will be defined as an absence of hypopigmentary changes and by a restoration of hyperpigmentary changes to mild or less at 6 month. Photographs of treated skin at follow-up visits will be compared to baseline to document the healing time course and may be used for blinded scoring evaluations (0-9 scales) of wrinkles, skin texture and color changes. The investigator will grade the epidermal response including side effects and adverse events using the 0 to 10 grading scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Kenkel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center Dept. of Plastic Surgery, Dallas, Texas, United States